CLINICAL TRIAL: NCT01964768
Title: Determination of Sensitivity and Specificity of Three Solutions of Allergen Extract (5 Grasses, Birch Pollens and Dermatophagoides Pteronyssinus Mites) for Diagnosis by Skin Prick Testing
Brief Title: Sensitivity and Specificity of 3 Solutions of Allergen Extract for Diagnosis by Skin Prick Testing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: DG40.08
Record Dates: First submitted 2013-10-10; First posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Patch Tests

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Skin prick-test

SUMMARY:
A Phase III study to determine the sensitivity and specificity of three solutions of different allergen extracts for diagnosis by skin prick-test:

* 5 Grasses pollen,
* Birch pollen,
* Dermatophagoides pteronyssinus mite

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study
* Male or female subjects aged 5-60 years inclusive
* Female of childbearing potential must be on a reliable method of contraception and have a negative urine pregnancy test
* Presence of a clinical history of allergy: seasonal or perennial rhinitis, conjunctivitis and/or asthma during grass or birch pollen seasons (at least two pollen seasons) and/or due to mite exposure (at least two years)
* Subjects affiliated to a social security system

Exclusion Criteria:

* Pregnant or breastfeeding women
* Dermographism
* Absence of cutaneous reactivity
* Presence of cutaneous lesions on the forearms either preventing the performance of the test or potentially interfering with the interpretation of the test
* Subjects presenting unstable asthma or poor general health condition
* Subjects with past or current specific immunotherapy treatment for any of the 3 tested allergens (Grass, Birch pollens, D. pteronyssinus and/or D. farinae mites) in the previous 5 years
* Any oral antihistaminic treatment in the previous 3 days or 10 days in case of loratadine or desloratadine
* Subjects on anti-IgE treatment
* Subjects treated with beta-blockers and/or anti-depressives.
* Subjects currently participating in another clinical trial or still in exclusion period for a previous clinical trial
* Investigators, co-investigators, as well as their children or spouses and all the study collaborators
* Subjects under protection of the courts, legal guardianship or legal trusteeship

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 324 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Skin wheal measure for each tested solution. For each allergen tested, 2 variables, positive SPT and negative SPT were defined. A SPT reaction was considered positive when the mean wheal diameter was >3 mm. A SPT reaction ≤3 mm was considered negative. | For each subject, the study consisted in one visit of about 60 minutes including skin prick-test and collection of blood sample for IgE determination.

SECONDARY OUTCOMES:
One of the secondary measurement was the wheal diameter for each allergen. | SPT measurements were performed after the study visit, an expected average of 1 week.

OTHER OUTCOMES:
The secondary measurement was also the specific IgE level for each allergen. | Specific IgE results were known after the study visit, an expected average of 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric de Blay, Pr, Principal Investigator — Hôpitaux Universitaires de Strasbourg, Nouvel Hôpital Civil, Strasbourg, France